CLINICAL TRIAL: NCT06518122
Title: A Randomized, Open Label, Multiple Dose, Crossover Clinical Trial to Evaluate the Drug-drug Interaction and Safety Between HCP1306, RLD2302 and RLD2102 in Healthy Volunteers
Brief Title: A Study to Evaluate the Drug-drug Interaction and Safety Between HCP1306, RLD2302 and RLD2102 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ROEM-101
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: [PART A] 6 x 3 Crossover
  [PART B] Single Arm (Three periods)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- [PART A] Sequence 1 (Experimental): Period1 : Treatment A (HCP1306) Period2 : Treatment B (RLD2302) Period3 : Treatment C (HCP1306+RLD2302)
  Interventions: Drug: HCP1306; Drug: RLD2302
- [PART A] Sequence 2 (Experimental): Period1 : Treatment C (HCP1306+RLD2302) Period2 : Treatment A (HCP1306) Period3 : Treatment B (RLD2302)
  Interventions: Drug: HCP1306; Drug: RLD2302
- [PART A] Sequence 3 (Experimental): Period1 : Treatment B (RLD2302) Period2 : Treatment C (HCP1306+RLD2302) Period3 : Treatment A (HCP1306)
  Interventions: Drug: HCP1306; Drug: RLD2302
- [PART A] Sequence 4 (Experimental): Period1 : Treatment C (HCP1306+RLD2302) Period2 : Treatment B (RLD2302) Period3 : Treatment A (HCP1306)
  Interventions: Drug: HCP1306; Drug: RLD2302
- [PART A] Sequence 5 (Experimental): Period1 : Treatment B (RLD2302) Period2 : Treatment A (HCP1306) Period3 : Treatment C (HCP1306+RLD2302)
  Interventions: Drug: HCP1306; Drug: RLD2302
- [PART A] Sequence 6 (Experimental): Period1 : Treatment A (HCP1306) Period2 : Treatment C (HCP1306+RLD2302) Period3 : Treatment B (RLD2302)
  Interventions: Drug: HCP1306; Drug: RLD2302
- [PART B] Single arm (Experimental): Period1 : Treatment D (RLD2102) Period2 : Treatment C (HCP1306) Period3 : Treatment E (HCP1306, RLD2302, RLD2102)
  Interventions: Drug: HCP1306; Drug: RLD2302; Drug: RLD2102

INTERVENTIONS:
Drug: HCP1306 — Take it once a day per period.
Drug: RLD2302 — Take it once a day per period.
Drug: RLD2102 — Take it once a day per period
  Arms: [PART B] Single arm

SUMMARY:
The purpose of this study is to evaluate the drug-drug interaction and safety between HCP1306, RLD2302 and RLD2102 in healthy volunteers.

DETAILED DESCRIPTION:
[PART A] To evaluate the drug-drug interaction and safety between HCP1306, RLD2302

[PART B] To evaluate the drug-drug interaction and safety between HCP1306, RLD2302, RLD2102

ELIGIBILITY:
Inclusion Criteria:

* Age 19~54 years in healthy volunteers
* 18.5 kg/m^2 ≤ BMI < 30 kg/m^2, weight(men) ≥55kg / weight(women) ≥45kg
* 90 mmHg ≤ SBP <140 mmHg, 50 mmHg ≤ DBP <90 mmHg
* Agrees that the person, spouse, or partner uses appropriate medically recognized contraception and does not provide sperm or eggs from the date of administration of the first investigational drug to 7 days after the administration of the last investigational drug
* Subjects who voluntarily decides to participate in this clinical trial and agree in writing to ensure compliance with the clinical trial

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
* Subjects who judged ineligible by the investigator

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
AUCtau | [PART A] 0~72 hours, [PART B] 0~48hours after final dose administration
  Pharmacokinetic evaluation
Css,max | [PART A] 0~72 hours, [PART B] 0~48hours after final dose administration
  Pharmacokinetic evaluation

SECONDARY OUTCOMES:
Css,min | [PART A] 0~72 hours, [PART B] 0~48hours after final dose administration
  Pharmacokinetic evaluation
Css,av | [PART A] 0~72 hours, [PART B] 0~48hours after final dose administration
  Pharmacokinetic evaluation
Tss,max | [PART A] 0~72 hours, [PART B] 0~48hours after final dose administration
  Pharmacokinetic evaluation
t1/2 | [PART A] 0~72 hours, [PART B] 0~48hours after final dose administration
  Pharmacokinetic evaluation
CLss/F | [PART A] 0~72 hours, [PART B] 0~48hours after final dose administration
  Pharmacokinetic evaluation
Vdss/F | [PART A] 0~72 hours, [PART B] 0~48hours after final dose administration
  Pharmacokinetic evaluation
Fluctuation[(Css,max-Css,min)/Css,av] | [PART A] 0~72 hours, [PART B] 0~48hours after final dose administration
  Pharmacokinetic evaluation
Swing[(Css,max-Css,min)/Css,min] | [PART A] 0~72 hours, [PART B] 0~48hours after final dose administration
  Pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Min-gul Kim, MD, Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Jeonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No